CLINICAL TRIAL: NCT05829421
Title: Feasibility of a Neuropsychologically Informed Occupational Therapy Intervention Targeting Decreased Ability to Perform Activities of Daily Living in People With Poststroke Cognitive Impairment
Brief Title: Addressing Problems in Managing Daily Tasks Due to Poststroke Cognitive Impairments
Acronym: NIOTI-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emma Ghaziani (Other)
Collaborators: Rigshospitalet, Denmark (Other); The Day Rehabilitation Centre, Frederiksberg Municipality, Denmark (Unknown); The Inpatient Rehabilitation Centre, Frederiksberg Municipality, Denmark (Unknown); Neurorehabilitation Centre Østervang, Frederiksberg Municipality, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Emma Ghaziani, Postdoc, OT, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-22066840
Record Dates: First submitted 2023-03-06; First posted 2023-04-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Impairment; Stroke
Keywords: occupational therapy; neuropsychology; stroke rehabilitation; cognitive rehabilitation; activities of daily living (ADL)
MeSH Terms: conditions — Cognitive Dysfunction; Stroke | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Feasibility study, non-randomised. An adaptive approach will be used to optimise the intervention content and study conduct as feasibility data are cumulated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impairment-specific occupational therapy (OT) intervention (Experimental): Patients receive an impairment-specific OT intervention targetting problems in managing activities of daily living (ADL) due to mild-to-moderate poststroke cognitive impairments. The intervention is initiated in the stroke unit as soon as patients' medical condition allows it, and it is delivered 3 times per week until 3 months poststroke. After hospital discharge, the intervention continues in community settings.
  Interventions: Other: Impairment-specific occupational therapy (OT) intervention

INTERVENTIONS:
Other: Impairment-specific occupational therapy (OT) intervention — In parallel with standard practice, patients receive an OT intervention adapted to the specific underlying cognitive impairments that are likely to disturb their performance of ADLs.
  The intervention is individualised through a 3-step process: a) a list of dysfunctional ADL process skills is forwarded by the OT to the neuropsychologist (NP), b) the NP identifies the cognitive impairments which are most likely to cause the dysfunctional ADL process skills through a cognitive assessment, c) based on the identified cognitive impairments, the NP and the OT select in collaboration the cognitive strategies that are most likely to benefit the individual patient from a pre-prepared intervention manual. Because of the large heterogeneity in how cognitive impairments impact on ADL performance, the exact way of implementing the selected cognitive strategies into the practice of the individual patient is left to the OT´s clinical judgement.

SUMMARY:
The purpose of this study is to investigate feasibility aspects of an intervention targeting problems in managing daily tasks due to mild-to-moderate poststroke cognitive impairments. We will specifically address uncertainties related to intervention content and delivery, and trial design and conduct.

ELIGIBILITY:
PATIENTS:

Inclusion criteria:

* first-ever symptomatic stroke,
* age ≥ 18 years,
* residence in Frederiksberg Municipality, Denmark,
* independent in pre-stroke everyday life (≤ 2 points on the modified Rankin Scale, mRS),
* experiencing problems in performing ADLs due to cognitive impairment; these problems are expected to still be present at hospital discharge,
* medical condition allows commencement of rehabilitation focused on ADL and cognition
* fully aware or mild-to-moderate unawareness of deficits (≤ 2 points on the Bisiach Anosognosia Scale, BAS),
* a global cognitive function corresponding to ≥ 17 points on the Montreal Cognitive Assessment, MoCA,
* ≤ 10 points on the depression subscale of the Hospital Anxiety and Depression Scale, HADS,
* able to provide informed consent, as evaluated by the recruiting healthcare professional(s),
* logistically possible to perform baseline assessments and create an individualised intervention plan during hospital stay
* provides informed consent

Exclusion criteria:

* psychiatric conditions causing difficulties or preventing participation, as evaluated by the recruiting health care professional(s)
* communication problems causing difficulties or preventing participation, as evaluated by the recruiting healthcare professional(s)

CAREGIVERS:

Inclusion criteria:

* appointed as close carer (by a patient who consented to participate),
* age ≥18y,
* provides informed consent.

Exclusion criteria:

-communication problems or other issues causing difficulties in participation as evaluated by the recruiting healthcare professional(s).

Patients without a close carer will not be excluded.

CLINICAL STAFF:

Inclusion criteria:

* appointed as local project managers, or OTs or NPs who conduct assessments or deliver the intervention in the participating centres,
* provides informed consent.

Exclusion criteria:

- unable to to follow a preliminary English version of the intervention manual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ADL process skills level (assessed by the Assessment of Motor and Process Skills, AMPS) at 3 months poststroke | At baseline (as soon as possible after stroke onset - expected:1 week poststroke) and 3 months poststroke
  The AMPS is a standardised observation-based instrument measuring two aspects of ADL performance: ADL motor skills (reflecting physical effort) and ADL process skills (reflecting efficiency, safety, and independence). The quality of each skill is evaluated on a 4-level scale. Based on Rasch statistics, the AMPS software converts these raw scores into two overall linear ADL scores (expressed in logits): an ADL motor score, and an ADL process score. Several studies support the AMPS' validity and reliability in both stroke populations. The AMPS is an OT-specific instrument and requires user certification.

SECONDARY OUTCOMES:
Change from baseline in ADL motor skills level (assessed by the Assessment of Motor and Process Skills, AMPS) at 3 months poststroke | At baseline (as soon as possible after stroke onset - expected:1 week poststroke) and 3 months poststroke
  The AMPS is a standardised observation-based instrument measuring two aspects of ADL performance: ADL motor skills (reflecting physical effort) and ADL process skills (reflecting efficiency, safety, and independence). The quality of each skill is evaluated on a 4-level scale. Based on Rasch statistics, the AMPS software converts these raw scores into two overall linear ADL scores (expressed in logits): an ADL motor score, and an ADL process score. Several studies support the AMPS' validity and reliability in both stroke populations. The AMPS is an OT-specific instrument and requires user certification.
Change from pre-stroke in global disability (assessed by the modified Rankin Scale, mRS) at 3 months. Min-max values: 0 (no symptoms at all) - 6 (dead) | At baseline (as soon as possible after stroke onset - expected:1 week poststroke) and 3 months poststroke
  Stroke-specific measure of global disability. Min-max values: 0 (no symptoms at all9 - 6 (dead).
Patient perceived health-related quality of life (assessed by the EuroQol-5D-5L, EQ-5D-5L) at 3 months poststroke | At 3 months poststroke
  Generic measure of health-related quality of life. It contains six subscales: mobility, self-care, usual activities, pain/discomfort, anxiety depression and perceived health. Perceived health is measured on a 0-100 scale (0: worst outcome, 100: best outcome). Each of remaining subscales are scored on a 5-level ordinal scale (1: best outcome, 5: worse outcome). The result for each subscale will be presented separately.
Caregiver perceived burden of stroke (assessed by the Caregiver Burden Scale, CBS) at 3 months posttsroke. | At 3 months poststroke
  The CBS is a 22-item scale that assess subjectively experienced burden by caregiver's to chronically disabled persons.
  The caregiver is asked to tick one of the four boxes (not at all, seldom, sometimes, often) score 1 to 4 for each question.
  The instrument comprises five factors: general strain, isolation, disappointment, emotional involvement and environment.
  A mean value is calculated for each factor including the following items:
  General strain: 1, 3, 4, 5, 7, 10, 14, and 19 Isolation: 8, 12, and 22 Disappointment: 2, 13, 18, 20, and 21 Emotional involvement: 6, 11, and 16 Environment: 9, 15, and 17

OTHER OUTCOMES:
Forms collecting feedback from project staff | Through study completion, an average of 1 year
  Based on feedback from the project staff collected through forms, the investigators will explore feasibility aspects such as: OTs' acceptability of the intervention, piloting the individualisation of the intervention, piloting the intervention delivery, refining the intervention manual, estimating participant recruitment and retention for a future RCT, and piloting outcome measures. .
Work meetings collecting feedback from project staff | Through study completion, an average of 1 year
  Based on feedback from the project staff collected through work meetings, the investigators will explore feasibility aspects such as: OTs' acceptability of the intervention, piloting the individualisation of the intervention, piloting the intervention delivery, and refining the intervention manual.
Semi-structured interviews collecting feedback from patient and caregivers | Through study completion, an average of 1 year
  Based on feedback from patients and caregivers, the investigators will explore the patients' acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Christensen, Professor, Principal Investigator — Bispebjerg and Frederiksberg Hospital
Locations (4):
- Denmark (4):
  - Bispebjerg and Frederiksberg Hospital, Copenhagen
  - Neurorehabilitation Centre Østervang, Frederiksberg
  - the Day Rehabilitation Centre, Frederiksberg
  - the Inpatient Rehabilitation Centre, Frederiksberg

IPD SHARING:
Plan to Share IPD: No